CLINICAL TRIAL: NCT01121432
Title: Diagnosis of Mediastinal Tuberculous Lymphadenopathy by Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chao-Chi Ho, National Taiwan University Hospital
Other Study IDs: 201003061R
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-04

CONDITIONS: Mediastinal Lymphadenopathy; Tuberculous Mediastinal Lymphadenopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mediastinal lymph nodes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mediastinal lymphadenopathy
  Interventions: Procedure: endobronchial ultrasound-guided transbronchial needle aspiration

INTERVENTIONS:
Procedure: endobronchial ultrasound-guided transbronchial needle aspiration — One time for aspiration/biopsy. The duration about 1-2 hour.

SUMMARY:
Although mediastinal tuberculous lymphadenopathy is not rare in adults of such an abnormality. Isolated mediastinal without a parenchymal lung lesion in adults is unusual with the incidence of 0.25%-5.8%. It occurs most commonly in Asian and black people, and presents a diagnostic problem. The definite diagnosis requires microbiology or pathology study.

Cervical mediastinoscopy remained the gold standard to sample the mediastnial lymph nodes, but this technique can access lymph node station 1-4, 7 only. EBUS-TBNA allows the mediastinal lymph nodes to be targeted in the areas accessible to cervical mediastinoscopy, as well as some hilar nodes (lymph node stations 2-4, 7, 10-12). Currently, the main indication of EBUS-TBNA is the mediastinal nodal staging of NSCLC after recent meta-analyses established the comparable sensitivity and specificity of nodal staging by EBUS-TBNA and cervical mediastinoscopy. Theoretically, mediastnial tuberculous lymphadenopathy could be diagnosed by the method of EBUS-TBNA. Douglas F. Johnson was the first doctor to report 2 cases of mediastinal tuberculous lymphadenopathy diagnosed by EBUS-TBNA in 2009. There are currently no much data on the use of this technique in this field. The investigators plan to perform a prospective single-center study to investigate the diagnostic efficacy of mediastinal tuberculous lymphadenopathy by sampling the culprit nodes via EBUS-TBNA. Concomitant sputum specimen for acid-fast stain and mycobacterial culture were collected as well.

DETAILED DESCRIPTION:
Although mediastinal tuberculous lymphadenopathy is much more common as a manifestation of primary tuberculosis in children, the presentation in adults of such an abnormality is not rare. In a large series reported in 1959 by Lyons and coworkers, tuberculosis was the 5th commonest cause of mediastinal enlargement, accounting for 6% of 782 cases. Intrathoracic lymphadenitis had been found to be present in between 0.5% and 26%.

However, isolated mediastinal without a parenchymal lung lesion in adults is unusual with the incidence of 0.25%-5.8%. It occurs most commonly in Asian and black people, and presents a diagnostic problem. Although chest CT findings such as nodes with central low attenuation and peripheral rim enhancement are suggestive, the definite diagnosis requires microbiology or pathology study.

Cervical mediastinoscopy remained the gold standard to sample the mediastnial lymph nodes, but this technique can access lymph node station 1-4, 7 only. EBUS-TBNA allows the mediastinal lymph nodes to be targeted in the areas accessible to cervical mediastinoscopy, as well as some hilar nodes (lymph node stations 2-4, 7, 10-12).

Kazuhiro Yasufuku had published the first report of rear-time EBUS-TBNA in evaluating mediastinal lymphadenopathy in 2004. Currently, the main indication of EBUS-TBNA is the mediastinal nodal staging of NSCLC after recent meta-analyses established the comparable sensitivity and specificity of nodal staging by EBUS-TBNA and cervical mediastinoscopy. Efficacy in evaluation of other disease processes such as sarcoidosis and lymphoma has also been established.

Theoretically, mediastnial tuberculous lymphadenopathy could be diagnosed by the method of EBUS-TBNA. Douglas F. Johnson was the first doctor to report 2 cases of mediastinal tuberculous lymphadenopathy diagnosed by EBUS-TBNA in 2009. There are currently no much data on the use of this technique in this field.

We plan to perform a prospective single-center study to investigate the diagnostic efficacy of mediastinal tuberculous lymphadenopathy by sampling the culprit nodes via EBUS-TBNA. Concomitant sputum specimen for acid-fast stain and mycobacterial culture were collected as well.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with mediastinal lymphadenopathy of unknown etiology
2. All patients signed informed consent before the procedure.

Exclusion Criteria:

1. Age less than 18 years
2. Bleeding diathesis (INR>1.4 or platelet count<10k/mcl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with mediastinal lymphadenopathy of unknow etiology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The ratio of tuberculous mediastinal lymphadenopathy | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan